CLINICAL TRIAL: NCT02297776
Title: Circulating Biomarkers Predict Neurological Outcome After Cardiac Arrest
Acronym: CABNO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Chen Yuanzhuo, M.D., Shanghai 10th People's Hospital
Other Study IDs: 040114001
Record Dates: First submitted 2014-11-16; First posted 2014-11-21 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; biomarker; microRNA; circRNA; NSE; CPC
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples are to be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CPC score 1 to 2: The patients with CPC score 1 to 2 judged half a year after cardiac arrest
- CPC scores 3 to 5: The patients with CPC score 3 to 5 judged half a year after cardiac arrest

SUMMARY:
Prediction of clinical outcome after cardiac arrest is clinically important.Early prognostication after successful cardiopulmonary resuscitation is difficult, and there is a need for novel methods to estimate the extent of brain injury and predict outcome. In this study, the investigators will evaluate the plasma levels of microRNAs (miRNAs) and circRNAs after cardiac arrest and assessed their ability to prognosticate neurological outcome.

DETAILED DESCRIPTION:
1. Diagnostic criteria for cardiac arrest Sudden loss of consciousness, carotid or femoral artery pulse disappeared, ECG showed ventricular asystole or ventricular fibrillation or ventricular tachycardia.
2. Diagnostic criteria for ROSC Recovery of complexion, autonomous aorta pulse can be detected, blood pressure> 90/60 mmHg, the condition above maintained stable for more than half an hour, defined as ROSC, otherwise as failed.
3. Clinical treatment CPR was applied according to the AHA2010 guidelines. Patients were admitted to SICU or EICU after confirmation of ROSC, and physical cooling machines were set at 33 degrees Celsius to protect brain within 24h after ROSC. Standard treatments for life support were performed for all the included patients.
4. Methods 4.1 Clinical data Data such as patient's age, gender, contact information, previous disease information, the major reason causing cardiac arrest, initial rhythm, the total time of CPR, utilization of an automatic chest compression device, time from cardiac arrest to ROSC and time from cardiac arrest to ICU admission was collected from each patient who was included in the study. Follow-up data for APARCHE II (acute physiology and chronic health evaluation scoring system) score, survival of 24 hours after cardiac arrest, survival of 48 hours after cardiac arrest, survival of 28 days after admission, CPC score 2 weeks after cardiac arrest and CPC score 6 months after cardiac arrest were collected.

4.2 Cerebral Performance Category (CPC) CPC is a 5-category scale for measuring neurological status 2 weeks after cardiac arrest and CPC score 6 months after cardiac arrest. The 5 categories are: CPC 1, conscious and alert with good cerebral performance; CPC 2, conscious and alert with moderate cerebral performance; CPC 3, conscious with severe cerebral disability; CPC 4, comatose or in persistent vegetative state; and CPC 5, brain dead, circulation preserved.

4.3 Sample collection and processing Whole blood sample was collected into Ethylene diamine tetra-acetic acid (EDTA) -anticoagulant tube from each patient immediately at the beginning of CPR, 24h, 48h and 7 days after cardiac arrest. Samples were centrifugated and the supernatant was stored in EP tube with out RNA enzyme at -80 degree Celsius.

4.4 Detection of miRNA and circRNA Patients were divided into two groups according to the Cerebral Performance Category （CPC） after half a year, "CPC 1-2 Group" and "CPC 3-5 Group". Five samples for 48h time point in each group were randomly selected and detected miRNA and circRNA with chips.The real-time quantitative PCR were used to detect the quantity of the selected miRNAs and circRNAs for each time point. The plasma concentration of NSE for each time point was tested by laboratory department.

ELIGIBILITY:
1 Inclusion criteria:

1. Transferred to or hospitalized in the emergency department or other wards of Shanghai Tenth People's Hospital due to cardiac arrest;
2. Return of spontaneous circulation (ROSC)after cardiopulmonary resuscitation;
3. Age > 14 years and < 85 years;
4. Written informed consent was obtained from all patients'family members before entering the study.

2 Exclusion criteria:

1. No witnesses when cardiac arrest occurs;
2. Obvious neurological dysfunction prior to cardiac arrest;
3. Intracranial infection or cerebrovascular accidents as primary disease or secondary complication within six months in the follow-up period.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: transferred to or hospitalized in the emergency department or other wards of Shanghai Tenth People's Hospital due to cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
cerebral performance Category（CPC) of Participants | up to 6 months after cardiopulmonary resuscitation

SECONDARY OUTCOMES:
survival of participants | up to 28 days after hospitalization
cerebral performance Category（CPC) of Participants | up to 2 weeks after cardiopulmonary resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Yuanzhuo Chen, MD, Study Chair — Shanghai 10th People's Hospital; Wenjie Li, MD, Principal Investigator — Shanghai 10th People's Hospital; Huiqi Wang, MD, Principal Investigator — Shanghai 10th People's Hospital; Chengjin Gao, MD, Study Director — Shanghai 10th People's Hospital; Hu Peng, MD, Study Director — Shanghai 10th People's Hospital; Yugang Zhuang, MD, Principal Investigator — Shanghai 10th People's Hospital; Xiangyu Zhang, MD, Study Director — Shanghai 10th People's Hospital; Qixing Wang, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth Hospital, Shanghai, China

REFERENCES:
- [Derived] Zhuang YG, Chen YZ, Zhou SQ, Peng H, Chen YQ, Li DJ. High plasma levels of pro-inflammatory factors interleukin-17 and interleukin-23 are associated with poor outcome of cardiac-arrest patients: a single center experience. BMC Cardiovasc Disord. 2020 Apr 15;20(1):170. doi: 10.1186/s12872-020-01451-y. PMID 32293300